CLINICAL TRIAL: NCT07362290
Title: TSPO Occupancy in the Human Lung
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 24/YH/0091
Record Dates: First submitted 2025-09-30; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Healthy Volunteers - Male and Female
MeSH Terms: interventions — N-benzyl-N-ethyl-2-(7,8-dihydro-7-methyl-8-oxo-2-phenyl-9H-purin-9-yl)acetamide

STUDY DESIGN:
Intervention Model Description: Part A will look at the TSPO signal in the lungs of participants, in the presence and absence of a drug to block the specific binding of the PET signal (XBD173). Part B will look at plasma concentrations of XBD173 following oral dosing (in fasting and fed states). This is a single group assignment where participants can take part in both Part A and Part B, or Part A alone, or Part B alone. Parts A and B will run concurrently
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The TSPO signal in the lungs of healthy individuals, in the presence and absence of XBD173 (Other): In part A, the investigators will use positron emission tomography (PET) imaging with the TSPO targeting PET ligand [11C]PBR28 to quantify the amount of TSPO in the lung. The investigators will then administer XBD173 orally (between 10mg and 90mg), and perform two subsequent [11C]PBR28 PET scans spread between two and 24 hours post dosing. XBD173 and [11C]PBR28 both bind the same site on the TSPO, and therefore compete with each other for TSPO binding. This allows for quantification of TSPO occupancy by XBD173. Measuring XBD173 plasma concentrations during the PET scan will allow us to learn how much XBD173 is required in the plasma to produce a certain degree of TSPO occupancy in the lung. Using a wide range of doses (10mg-90mg) and scan times (2-24 hours) ensures that some participants will have high TSPO occupancy and some will have low TSPO occupancy. This will allow us to better understand the plasma concentration/occupancy relationship.
  Interventions: Drug: XBD173
- Plasma concentrations of XBD173 following oral dosing (in fasting and fed states) (Other): Part B will look at what doses of XBD173 are required to achieve the plasma concentration leading to high TSPO occupancy at steady state (to be determined in Part A), and whether taking XBD173 with food affects the plasma concentrations achieved. The investigatorsassume that the plasma concentrations required to cause high TSPO occupancy (identified in Part A) will be achieved with a dose of approximately 60mg. Therefore, in Part B for study visits 1, 2 and 3, participants will receive 6 doses of 60mg XBD173 spread over 3 days and the effect of food investigated by dosing with and without food.
  Interventions: Drug: XBD173

INTERVENTIONS:
Drug: XBD173 — Small molecule experimental medication binding to mitochondrial protein TSPO

SUMMARY:
The investigators would like to explore the role of TSPO in PAH using a pharmacological challenge agent (XBD173) to modulate TSPO function. In order to appropriately design experimental medicine studies examining TSPO function, the investigators first need an understanding of the relationship between XBD173 dose and occupancy of lung TSPO.

The aim of the proposed study, therefore, is to answer three questions:

1. What plasma concentrations of XBD173 are required to cause high occupancy of lung TSPO?
2. What doses of XBD173 are required to achieve these plasma concentrations at steady state?
3. Does taking XBD173 with food affect the plasma concentrations achieved?

Part A will address question (1). In part A, the investigators will use positron emission tomography (PET) imaging with the TSPO targeting PET ligand [11C]PBR28 to quantify the amount of TSPO in the lung. The investigators will then administer XBD173 orally (between 10mg and 90mg), and perform two subsequent [11C]PBR28 PET scans. XBD173 and [11C]PBR28 both bind the same site on the TSPO, and therefore compete with each other for TSPO binding. This allows for quantification of TSPO occupancy by XBD173. Measuring XBD173 plasma concentrations during the PET scan will allow the investigators to learn how much XBD173 is required in the plasma to produce a certain degree of TSPO occupancy in the lung. Using a wide range of doses (10mg-90mg) and scan times ensures that some participants will have high TSPO occupancy and some will have low TSPO occupancy. This will allow the investigators to better understand the plasma concentration/occupancy relationship.

Part B will address questions (2) and (3), i.e what doses of XBD173 are required to achieve the plasma concentration leading to high TSPO occupancy at steady state (to be determined in Part A), and does taking XBD173 with food affect the plasma concentrations achieved? The investigators assume that the plasma concentrations required to cause high TSPO occupancy (identified in Part A) will be achieved with a dose of approximately 60mg. Therefore, in Part B for study visits 1, 2 and 3, participants will receive 6 doses of 60mg XBD173 spread over 3 days and the effect of food investigated by dosing with and without food.

In Part A at Study Visit 1, a [11C]-PBR28 PET scan will be performed under baseline conditions. XBD173 will then be administered (10-90mg, oral) on study visits 2 and 3 and two further PET scans will be performed post dosing to understand how long the drug blocks the binding of the PET tracer.

The first two participants will be dosed with 10-90mg. The dose and scan times for remaining subjects will be based on occupancy and plasma drug level data for previous subjects.

In Part B at Study Visit 1, participants will arrive fasted in the morning. After placement of a venous cannula will then be dosed with a single dose of oral XBD173 (60mg). Blood samples will be taken at up to 12 timepoints over 8 hours. At Study Visit 2, participants will arrive fasted in the morning. They will be given a standard breakfast and the procedures of Study Visit 1 will be repeated, with dosing occurring within 15 mins of finishing breakfast. They will receive a second dose of XBD173 (60mg) whilst at the ICRF 6-8 hours after the first dose, having had lunch. Participants will then be given a further dose to take at home that night prior to bed. At Study Visit 3, which will occur on the following day, participants will arrive in the morning fasted and will be given a standard breakfast. After placement of a venous cannula, they will be dosed orally with XBD173 (60mg) in the morning and again 6-8 hours later, and blood samples taken throughout the day.

Study visits 4, 5 and 6 will be identical to Study visits 1,2 and 3 respectively, but for the dose of XBD173 which will be 40mg or 90mg depending on the plasma levels obtained with 60mg.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged between 25-75 years old
* Able to provide written informed consent prior to any study mandated procedures
* Able to lie comfortably on back for up to 90 minutes at a time (Part A only)
* Female participants of childbearing potential are eligible to participate after a negative highly sensitive pregnancy test if they are taking a highly effective method of contraception during participation in the study and until the end of relevant systemic exposure. The following methods are permitted:
* progesterone implant
* intrauterine device (also called IUD)
* intrauterine hormone-releasing system (also known as IUS)
* bilateral tubal occlusion
* vasectomised partner
* sexual abstinence
* Male participants who are fertile are eligible to participate if they are willing to comply with the contraceptive requirements as listed above *Definition of fertile females (women of childbearing potential) and of fertile men: For the purpose of this document, a woman is considered of childbearing potential, i.e. fertile, following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilisation methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy. A postmenopausal state is defined as no menses for 12 months without an alternative medical cause. A high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a post-menopausal state in women not using hormonal contraception or hormonal replacement therapy. However in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient. For the purpose of this document, a man is considered fertile after puberty unless their medical notes document that they are permanently sterile.

Exclusion Criteria:

* Unable to provide informed consent and/or are non-fluent speakers of the English language
* Hypersensitivity to XBD173 or to any of the excipients
* Clinically-significant renal disease (confirmed by creatinine clearance <30 ml/min per 1.73m2)
* Clinically-significant liver disease (confirmed by serum transaminases >3 times than upper normal limit)
* History of uncontrolled systemic hypertension
* Acute infection (including eye, dental, and skin infections)
* History of chronic inflammatory disease including HIV, and Hepatitis B
* Women who are pregnant or breastfeeding
* Patients who have received an Investigational Medicinal Product (IMP) within 5 half-lives of the last dose of the IMP or 1 month (which ever is greater) before the baseline visit
* Diagnosis of any condition which may directly or indirectly lead to lung pathology in the opinion of the investigator
* Severe and moderate P450 CY3A4 inhibitors

  o Boceprevir, Clarithromycin, Cobicistat, Idelalisib, Itraconazole, Ketoconazole, Nelfinavir, Ritonavir, Saquinavir, Telaprevir, Telithromycin, Voriconazoleb, Aprepitant, Conivaptan, Crizotinib, Diltiazem, Dronedarone, Erythromycin, Fluconazole, Imatinib, Isavuconazole, Nefazodone, Netupitant, Nilotinib, Posaconazolee, Tofisopam, Verapamil, Delavirdine.
* Severe and moderate P450 CY3A4 inducers

  o Carbamazepine, Enzalutamide, Fosphenytoin, Mitotane, Phenytoin, Rifampicin, Bosentan, Efavirenz, St John's wort, Barbiturates, Nevirapine, Primidone, Rifabutin, Rifapentine.
* Part A (PET imaging) specific exclusion criteria

  * TT/AT Genotype at the rs6971 locus
  * Previous participation in a research study involving ionising radiation such that in combination with this study the radiation exposure over the last 12 months would exceed 10 mSv
  * Positive Allen's test
  * Use of Oral anticoagulants or antiplatelet agents other than low dose aspirin

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-09-19 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
To establish the relationship between plasma concentration of XBD173 and TSPO occupancy in the human lung | Up to 4 months
  This will be achieved by measuring the [11C]PBR28 signal in the lungs of healthy individuals in the presence and absence of XBD173. We will use Occupancy % to measure this outcome. [11C]PBR28 signal in the lungs will be measured by volume of distribution.

SECONDARY OUTCOMES:
To establish the relationship between dose of XBD173 and plasma concentration of XBD173 at steady state , fed state and fasted state. | Up to 1 week
  This will be achieved by measuring the XBD173 plasma concentration at steady state, fed state and fasted state.

CONTACTS AND LOCATIONS:
Locations (1):
- NIHR Imperial CRF, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No